CLINICAL TRIAL: NCT05718284
Title: High Flow Nasal Cannula Oxygen Administration Versus Standard Care After Esophagectomy for Cancer: a Randomized Controlled Trial.
Brief Title: High Flow Nasal Cannula After Esophagectomy
Acronym: OSSIGENA1V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cristian Deana (Other)
Responsible Party: Sponsor-Investigator, Cristian Deana, MEDICAL doctor, Anesthesiologist and Critical Care Physician, Azienda Sanitaria-Universitaria Integrata di Udine
Organization: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSSIGENA
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Cancer; Postoperative Pulmonary Atelectasis; Postoperative Pneumonia; Postoperative Pneumothorax; Postoperative Infection of Incision; Postoperative Acute Myocardial Infarction
Keywords: esophageal cancer; anesthesia; high flow nasal cannula; pneumonia; esophagectomy; acute myocardial infarction
MeSH Terms: conditions — Esophageal Neoplasms; Pulmonary Atelectasis; Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Experimental): Administration of high flow nasal oxygen after extubation for 48 hours
  Interventions: Device: AIRVO2
- STANDARD OXYGEN (Other): Administration of oxygen through standard devices (nasal cannulae, venturi mask, none)
  Interventions: Other: STANDARD CARE

INTERVENTIONS:
Device: AIRVO2 — APPLICATION OF HIGH FLOW NASAL CANNULA OXYGEN FOR 48 HOURS AFTER ESOPHAGECTOMY
  Arms: HFNC
Other: STANDARD CARE — APPLICATION OF OXYGEN THROUGH STANDARD CARE FOR 48 HOURS AFTER ESOPHAGECTOMY
  Arms: STANDARD OXYGEN

SUMMARY:
This study will compare the effect of HFNC versus standard oxygen administration after elective esophagectomy for cancer.

ELIGIBILITY:
Inclusion Criteria:

* elective esophagectomy for cancer
* METS≥4
* AGE 18-85
* Written informed consent

Exclusion Criteria:

* ASA>3
* COPD≥ III stage according to GOLD criteria
* FEV1<50%
* EF<30%
* NYHA>2
* BMI<17 or >35 Kg/m2
* CKD with eGFR<60 mL/min

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
POST-OPERATIVE PULMONARY COMPLICATIONS | within 30 days after surgery
  Describe the frequency of PPC that include: pneumonia, pleural effusion, pneumothorax, atelectasis, ARDS, aspiration pneumonia, trachea-bronchial lesion, air leak

SECONDARY OUTCOMES:
CARDIO-VASCULAR COMPLICATIONS | within 30 days after surgery
  Describe the frequency of myocardial infarction, pulmonary edema, cardiac arrest, pulmonary embolism, deep venous thrombosis, stroke, pericardtis

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Universitaria Friuli Centrale, Udine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deana C, Vetrugno L, Stefani F, Basso A, Matellon C, Barbariol F, Vecchiato M, Ziccarelli A, Valent F, Bove T, Bassi F, Petri R, De Monte A. Postoperative complications after minimally invasive esophagectomy in the prone position: any anesthesia-related factor? Tumori. 2021 Dec;107(6):525-535. doi: 10.1177/0300891620979358. Epub 2020 Dec 15. PMID 33323061
- [Background] Xia M, Li W, Yao J, Jin Y, Du G, Xu Q, Yi X, Nv X, Wu Y, He P, Wu W. A postoperative comparison of high-flow nasal cannula therapy and conventional oxygen therapy for esophageal cancer patients. Ann Palliat Med. 2021 Mar;10(3):2530-2539. doi: 10.21037/apm-20-1539. Epub 2021 Jan 21. PMID 33548991
- [Derived] Deana C, Vecchiato M, Azzolina D, Turi S, Boscolo A, Pistollato E, Skurzak S, Amici O, Priolo S, Tonini S, Foti LS, Taddei E, Aceto P, Martino A, Ziccarelli A, Cereser L, Andreutti S, De Carlo S, Lirussi K, Barbariol F, Cammarota G, Polati E, Forfori F, Corradi F, Patruno V, Navalesi P, Maggiore SM, Lucchese F, Petri R, Bassi F, Romagnoli S, Bignami EG, Vetrugno L; Ossigena Study Group. Effect on post-operative pulmonary complications frequency of high flow nasal oxygen versus standard oxygen therapy in patients undergoing esophagectomy for cancer: study protocol for a randomized controlled trial-OSSIGENA study. J Thorac Dis. 2024 Aug 31;16(8):5388-5398. doi: 10.21037/jtd-24-575. Epub 2024 Aug 13. PMID 39268119